CLINICAL TRIAL: NCT00325403
Title: A 12-Week, International, Multicenter, Double-Blind, Randomized, Placebo-Controlled Comparison of the Efficacy and Safety of Oral UT-15C Sustained Release Tablets in Subjects With Pulmonary Arterial Hypertension
Brief Title: FREEDOM - M: Oral Treprostinil as Monotherapy for the Treatment of Pulmonary Arterial Hypertension (PAH)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TDE-PH-302
Record Dates: First submitted 2006-05-11; First posted 2006-05-12 (Estimated); Results first posted 2013-03-18 (Estimated); Last update posted 2024-01-03 (Actual); Status verified 2013-02

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension | interventions — treprostinil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- UT-15C (oral treprositnil) (Active Comparator): Subjects receive UT-15C (oral treprostinil) twice daily.
  Interventions: Drug: Oral treprostinil (UT-15C) Sustained Release Tablets
- Placebo (Placebo Comparator): Subjects receive placebo (sugar pill) twice daily.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Oral treprostinil (UT-15C) Sustained Release Tablets — Sustained release oral tablet, twice daily
  Other Names: treprostinil diethanolamine
  Arms: UT-15C (oral treprositnil)
Other: Placebo — Placebo oral tablet twice daily
  Arms: Placebo

SUMMARY:
This study was an international, multicenter, randomized (2:1 active:placebo), double-blind, placebo-controlled study in subjects with PAH who were NOT currently receiving approved therapy for their PAH. Study visits occurred at 4 week intervals for 12 weeks (with an additional visit at Week 11) with the key measure of efficacy being the 6-minute walk test. Study procedures included routine blood tests, medical history, physical exams, disease evaluation, and exercise tests. Two optional substudies were also a part of FREEDOM-M at select centers - a hemodynamic substudy with a right heart catheterization at Baseline and Week 12 and a genetics and biomarkers substudy with blood samples collected at Baseline and Week 12.

Patients who completed all assessments for 12 weeks were also eligible to enter an open-label, extension phase study (FREEDOM - EXT).

ELIGIBILITY:
Inclusion Criteria:

* Between 12 and 75 years of age, inclusive.
* Body weight at least 40 kg with a Body Mass Index < 45
* PAH that is either idiopathic/heritable; associated with repaired congenital systemic-to-pulmonary shunts (repaired ≥ 5 years); associated with collagen vascular disease; associated with HIV.
* Previous testing (e.g., right heart catheterization, echocardiography) consistent with the diagnosis of PAH.
* Baseline 6-minute walk distance between 200 and 425 meters, inclusive.
* Reliable and cooperative with protocol requirements.

Exclusion Criteria:

* Nursing or pregnant.
* Currently receiving an endothelin receptor antagonist, a phosphodiesterase-5 inhibitor, or prostacyclin within 30 days of Baseline.
* PAH due to conditions other than noted in the above inclusion criteria.
* History of uncontrolled sleep apnea, renal insufficiency, anemia, left sided heart disease, uncontrolled systemic hypertension, or parenchymal lung disease.
* Use of an investigational drug within 30 days of Baseline.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2006-10; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Laliberte, PharmD, Study Director — United Therapeutics
Locations (77):
- United States (43):
  - University of Alabama-Birmingham, Birmingham, Alabama
  - Arizona Pulmonary Specialist, Phoenix, Arizona
  - Mayo Clinic Arizona, Phoenix, Arizona
  - University of California, San Francisco-Fresno, Fresno, California
  - West Los Angeles VA Healthcare Center, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - Harbor-UCLA Medical Center, Torrance, California
  - University of Colorado Health Science Center, Aurora, Colorado
  - University of Florida - Shands Hospital, Jacksonville, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Emory University Hospital, Atlanta, Georgia
  - University of Chicago Hospitals, Chicago, Illinois
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - Kentuckiana Pulmonary Associates, Louisville, Kentucky
  - Alexandria Cardiology Clinic, Alexandria, Louisiana
  - Maine Medical Center, Portland, Maine
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University Hospital, St Louis, Missouri
  - Nebraska Medical Center, Omaha, Nebraska
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Winthrop University Hospital, Mineola, New York
  - Columbia Presbyterian Medical Center, New York, New York
  - Mary M Parkes Center for Asthma, Allergy and Pulmonary Care - University of Rochester, Rochester, New York
  - The Lindner Center, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Legacy Clinic Northwest, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Southwestern, Dallas, Texas
  - Baylor College of Medicine, Pulmonary & Critical Care, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Heart Care Associates, Milwaukee, Wisconsin
- Universitaet Wien, Vienna, Austria
- Belgium (2):
  - Hospital Erasme, Brussels
  - University Hospital Gasthuisberg, Leuven
- Canada (3):
  - Peter Lougheed Centre, Calgary, Alberta
  - London Health Science Centre, London, Ontario
  - SMBD Jewish General Hospital, Montreal, Quebec
- China (3):
  - Beijing Shijitan Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Shanghai Pulmonary Hospital, Shanghai
- Hospital Antoine Beclere, Clamart, France
- India (12):
  - PRIME Hospitals, Hyderbad, Andhra Pradesh
  - Care Institute of Medical Science, Ahmedabad, Gujarat
  - Lifecare Institute of Medical Sciences & Research, Ahmedabad, Gujarat
  - Narayana Hrudayalaya Institute of Medical Sciences, Bangalore, Karnataka
  - Asian Heart Institute and Research Centre, Parel Mumbai, Maharashtra
  - Poona Hospital and Research Centre, Pune, Maharashtra
  - Sri Ramachandra Medical College, Chennai, Tamil Nadu
  - G. Kuppuswamy Naidu Memorial Hospital, Coimbatore, Tamil Nadu
  - K. S. Hospital, Chennai, Tamil Nadu
  - Sir Ganga Ram Hospital, New Delhi
  - Ruby Hall Clinic, Pune
  - Care Hospital, Visakhapatnam, Andra Pradesh
- Israel (3):
  - Hadassah Ein-Kerem Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Tel Hashomer Medical Center, Ramat Gan
- Universita degli Studi Bologna, Bologna, Italy
- Mexico (3):
  - Instituto Nacional de Cardiologia, Mexico City, Mexico City
  - Hospital Universitario UANL, Monterrey, Nuevo León
  - Unidad de Investigacion Clinica en Medicina (UDICEM), Monterrey
- VU Medisch Centrum (VUCM), Amsterdam, Netherlands
- Poland (3):
  - Krakowski Szpital Specjalistyczny im. (Kraków Specialist Hospital), Krakow
  - National Tuberculosis and Lung Disease Research Institute, Warsaw
  - Wojewódzki Szpital Specjalistyczny we Wroclawiu (Provincial Specialist Hospital in Wrocław), Wroclaw
- Auxilio Mutuo Hospital, Guaynabo, Puerto Rico

REFERENCES:
- [Derived] Jing ZC, Parikh K, Pulido T, Jerjes-Sanchez C, White RJ, Allen R, Torbicki A, Xu KF, Yehle D, Laliberte K, Arneson C, Rubin LJ. Efficacy and safety of oral treprostinil monotherapy for the treatment of pulmonary arterial hypertension: a randomized, controlled trial. Circulation. 2013 Feb 5;127(5):624-33. doi: 10.1161/CIRCULATIONAHA.112.124388. Epub 2013 Jan 10. PMID 23307827
- See also: FREEDOM Studies Website — http://www.pahstudy.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 349 subjects participated in the study from 24 October 2006 to 29 April 2011 at 52 of 77 sites across the United States, Puerto Rico, Canada, Europe, Israel, India, Mexico, and China. The primary endpoint was analyzed using the primary analysis population which included 228 subjects who had access to 0.25 mg tablets at the time of randomization.
Groups:
- Placebo: These subjects were randomly allocated to receive matching oral placebo twice daily (every 12 hours +/- 1 hour) and were included in the primary analysis population. Dose increases were made in the absence of dose-limiting drug-related AEs, to ensure the subject received the optimal clinical dose throughout the study.
- UT-15C (Oral Treprostinil): These subjects were randomly allocated to receive oral treprostinil twice daily (every 12 hours +/- 1 hour) and were included in the primary analysis population. Dose increases were made in the absence of dose-limiting drug-related AEs, to ensure the subject received the optimal clinical dose throughout the study.
Period: Overall Study
Arm/Group | Placebo | UT-15C (Oral Treprostinil)
Started | 116 | 233
Completed | 98 (98 subjects receiving placebo completed the study on study drug) | 182 (182 subjects receiving oral treprostinil completed the study on study drug)
Not Completed | 18 | 51

BASELINE CHARACTERISTICS:
Groups:
- Placebo: These subjects were randomly allocated to receive placebo twice daily and were included in the primary analysis population. Baseline measures are provided for the modified intention to treat (mITT) group, which includes subjects with access to 0.25 mg tablets at randomization (n=228).
- UT-15C (Oral Treprostinil): These subjects were randomly allocated to receive oral treprostinil twice daily and were included in the primary analysis population. Baseline measures are provided for the modified intention to treat (mITT) group, which includes subjects with access to 0.25 mg tablets at randomization (n=228).
- Total: Total of all reporting groups
Arm/Group | Placebo | UT-15C (Oral Treprostinil) | Total
Number analyzed (Participants) | 77 | 151 | 228
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 9 | 10
  Between 18 and 65 years | 69 | 141 | 210
  >=65 years | 7 | 1 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (13.5) | 37.8 (13.5) | 39.4 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 108 | 166
  Male | 19 | 43 | 62
PAH Etiology [Number; unit: participants]
  Idiopathic or heritable PAH | 56 | 114 | 170
  PAH associated w collagen vascular disease | 17 | 26 | 43
  PAH associated w repaired congenital heart defect | 3 | 10 | 13
  PAH associated w HIV infection | 1 | 1 | 2
Baseline Six Minute Walk Distance [Mean (Standard Deviation); unit: meters] | 327.6 (70.7) | 331.3 (64.9) | 330.0 (66.8)
WHO Functional Classification [Number; unit: participants] — Class I: PH without limitation of physical activity (PA); no undue dyspnea or fatigue, chest pain, or near syncope.
  Class II: PH resulting in slight limitation of PA; comfortable at rest; ordinary PA causes undue dyspnea or fatigue, chest pain or near syncope.
  Class III: PH resulting in marked limitation of PA; comfortable at rest; ordinary PA causes undue dyspnea or fatigue, chest pain, or near syncope.
  Class IV: PH with inability to carry out any PA without symptoms and signs of right heart failure. Dyspnea and/or fatigue may be present at rest. Discomfort is increased by any PA.
  participants
    WHO Class I | 1 | 1 | 2
    WHO Class II | 24 | 52 | 76
    WHO Class III | 52 | 98 | 150

OUTCOME MEASURES:

1. Primary Outcome: Six Minute Walk Distance (6MWD)
Description: Placebo corrected change in six minute walk distance (6MWD) from Baseline to Week 12, correlates with the historical clinical standard for assessing patient functional status in the treatment of PAH and is considered an objective measure of patient functional status by the American Thoracic Society (ATS).
  The six minute walk test was to be conducted 3 to 6 hours after the previous dose of study drug.
  The Hodges-Lehmann median difference between treatment groups was used to estimate the treatment effect on 6MWD from Baseline to Week 12. A rank-based methodology was used instead of parametric-based methodology to avoid statistical bias caused by extreme outliers resulting from the handling of data that are missing due to death or clinical worsening of PAH. It is a more robust estimator than the between-treatment difference in medians.
Time Frame: Baseline and Week 12
Population: Analyses were conducted using the modified intention to treat (mITT) group, which includes subjects with access to 0.25 mg tablets at randomization (n=228). All alpha was spent on this subgroup, thereby maintaining an overall type I error rate of 0.05. For sensitivity purposes, efficacy analyses were also performed on all enrolled subjects (n=349).
Measure: Median (Inter-Quartile Range); unit: meters
Groups:
- Placebo: These subjects were randomly allocated to receive placebo twice daily and were included in the primary analysis population.
- UT-15C (Oral Treprostinil): These subjects were randomly allocated to receive oral treprostinil twice daily and were included in the primary analysis population.
Arm/Group | Placebo | UT-15C (Oral Treprostinil)
Number analyzed (Participants) | 77 | 151
meters
  6MWD at Baseline | 339 [282 to 381] | 350 [283 to 386]
  6MWD at Week 12 | 343 [246 to 403] | 370 [300 to 418]
  Change in 6MWD from Baseline to Week 12 | -5 [-41 to 49] | 25 [-16 to 63]
Statistical Analysis 1: Comparison: Placebo vs UT-15C (Oral Treprostinil); Using an allocation ratio of 2:1 between oral treprostinil and placebo, a fixed sample size of approximately 195 subjects with access to 0.25 mg tablets at randomization would provide at least 90% power at a significance level of 0.01 (two-sided hypothesis) to detect a between-treatment difference in the change from Baseline to Week 12 in distance traversed during the 6-minute walk, assuming a true underlying treatment difference of 45 meters with a SD of 75 meters in both treatment groups; Test type: Superiority or Other; p = 0.0125, ANCOVA — P-Value; Hodges-Lehmann (H-L) = 23, 95% CI 2-sided [4 to 41]

2. Secondary Outcome: Six Minute Walk Distance (6MWD)
Description: Placebo corrected change in six minute walk distance (6MWD) from Baseline to Week 11, a time expected to correlate with trough treprostinil concentration.
  The six minute walk test was to be conducted 8 to 13 hours after the previous dose of study drug.
  The Hodges-Lehmann median difference between treatment groups was used to estimate the treatment effect on 6MWD from Baseline to Week 11. A rank-based methodology was used instead of parametric-based methodology to avoid statistical bias caused by extreme outliers resulting from the handling of data that are missing due to death or clinical worsening of PAH. It is a more robust estimator than the between-treatment difference in medians.
Time Frame: Baseline and Week 11
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | Placebo | UT-15C (Oral Treprostinil)
Number analyzed (Participants) | 77 | 151
meters
  6MWD at Baseline | 339 [282 to 381] | 350 [283 to 386]
  6MWD at Week 11 | 335 [254 to 400] | 350 [290 to 400]
  Change in 6MWD from Baseline to Week 11 | 0 [-54 to 36] | 8 [-25 to 50]
Statistical Analysis 1: Comparison: Placebo vs UT-15C (Oral Treprostinil); Test type: Superiority or Other; p = 0.0653, ANCOVA; Hodges-Lehmann (H-L) = 13, 95% CI 2-sided [-2 to 33]

3. Secondary Outcome: Six Minute Walk Distance (6MWD)
Description: Placebo corrected change in six minute walk distance (6MWD) from Baseline to Week 8, correlates with the historical clinical standard for assessing patient functional status in the treatment of PAH and is considered an objective measure of patient functional status by the American Thoracic Society (ATS).
  The six minute walk test was to be conducted 3 to 6 hours after the previous dose of study drug.
  The Hodges-Lehmann median difference between treatment groups was used to estimate the treatment effect on 6MWD from Baseline to Week 8. A rank-based methodology was used instead of parametric-based methodology to avoid statistical bias caused by extreme outliers resulting from the handling of data that are missing due to death or clinical worsening of PAH. It is a more robust estimator than the between-treatment difference in medians.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | Placebo | UT-15C (Oral Treprostinil)
Number analyzed (Participants) | 77 | 151
meters
  6MWD at Baseline | 339 [282 to 381] | 350 [283 to 386]
  6MWD at Week 8 | 347 [240 to 398] | 355 [300 to 408]
  Change in 6MWD from Baseline to Week 8 | 0 [-36 to 35] | 17 [-15 to 54]
Statistical Analysis 1: Comparison: Placebo vs UT-15C (Oral Treprostinil); Test type: Superiority or Other; p = 0.0307, ANCOVA; Hodges-Lehmann (H-L) = 17, 95% CI 2-sided [1 to 33]

4. Secondary Outcome: Six Minute Walk Distance (6MWD)
Description: Placebo corrected change in six minute walk distance (6MWD) from Baseline to Week 4, correlates with the historical clinical standard for assessing patient functional status in the treatment of PAH and is considered an objective measure of patient functional status by the American Thoracic Society (ATS).
  The six minute walk test was to be conducted 3 to 6 hours after the previous dose of study drug.
  The Hodges-Lehmann median difference between treatment groups was used to estimate the treatment effect on 6MWD from Baseline to Week 4. A rank-based methodology was used instead of parametric-based methodology to avoid statistical bias caused by extreme outliers resulting from the handling of data that are missing due to death or clinical worsening of PAH. It is a more robust estimator than the between-treatment difference in medians.
Time Frame: Baseline and Week 4
Population: Analyses were conducted using the modified intention to treat (mITT), which includes subjects who had access to 0.25 mg tablets at randomization (n=228). All alpha was spent on this subgroup, thereby maintaining an overall type I error rate of 0.05. For sensitivity purposes, efficacy analyses were also performed on all enrolled subjects (n=349).
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | Placebo | UT-15C (Oral Treprostinil)
Number analyzed (Participants) | 77 | 151
meters
  6MWD at Baseline | 339 [282 to 381] | 350 [283 to 386]
  6MWD at Week 4 | 350 [254 to 387] | 360 [285 to 400]
  Change in 6MWD from Baseline to Week 4 | 0 [-28 to 17] | 7 [-15 to 42]
Statistical Analysis 1: Comparison: Placebo vs UT-15C (Oral Treprostinil); Test type: Superiority or Other; p = 0.0518, ANCOVA; Hodges-Lehmann (H-L) = 12, 95% CI 2-sided [0 to 24]

5. Secondary Outcome: Clinical Worsening Assessment
Description: Definition of clinical worsening included patients who met at least one of the following criteria during the 12 weeks of the study:
  1. Death (all causes excluding accident)
  2. Transplantation or atrial septostomy
  3. Clinical deterioration as defined by:
     1. Hospitalization as a result of PAH, or
     2. greater than or equal to 20% decrease in 6MWD from Baseline (or too ill to walk) and a decrease in WHO functional class And
     3. Initiation of new PAH specific therapy (i.e., ERA, PDE5-I, prostacyclin)
Time Frame: Baseline and Week 12
Measure: Number; unit: participants
Arm/Group | Placebo | UT-15C (Oral Treprostinil)
Number analyzed (Participants) | 77 | 151
participants | 8 | 15
Statistical Analysis 1: Comparison: Placebo vs UT-15C (Oral Treprostinil); Test type: Superiority or Other; p = 1.000, Fisher Exact

6. Secondary Outcome: World Health Organization Functional Classification for PAH
Description: Class I: Patients with pulmonary hypertension but without resulting limitation of physical activity. Ordinary physical activity does not cause undue dyspnea or fatigue, chest pain, or near syncope.
  Class II: Patients with pulmonary hypertension resulting in slight limitation of physical activity. These patients are comfortable at rest, but ordinary physical activity causes undue dyspnea or fatigue, chest pain or near syncope.
  Class III: Patients with pulmonary hypertension resulting in marked limitation of physical activity. They are comfortable at rest. Ordinary activity causes undue dyspnea or fatigue, chest pain, or near syncope.
  Class IV: Patients with pulmonary hypertension with inability to carry out any physical activity without symptoms. These patients manifest signs of right heart failure. Dyspnea and/or fatigue may be present even at rest. Discomfort is increased by any physical activity.
Time Frame: Baseline and Week 12
Population: Subjects with a WHO functional classification assessment at Week 12.
Measure: Number; unit: participants
Arm/Group | Placebo | UT-15C (Oral Treprostinil)
Number analyzed (Participants) | 77 | 151
participants
  WHO Class I | 1 | 2
  WHO Class II | 29 | 59
  WHO Class III | 38 | 75
  WHO Class IV | 9 | 15
Statistical Analysis 1: Comparison: Placebo vs UT-15C (Oral Treprostinil); Test type: Superiority or Other; p = 0.7380, Wilcoxon rank sum test — In cases where the "value corresponding to overall poorest relative change" was imputed for walk distance, a value of "IV" was used for the WHO functional classification for PAH; Hodges-Lehmann (H-L) = 0, 95% CI 2-sided [0 to 0] — The values for the estimated parameter and 95% confidence interval were calculated

7. Secondary Outcome: Borg Dyspnea Score
Description: The Borg dyspnea score is a 10-point scale rating the maximum level of dyspnea experienced during the 6-minute walk test. The Borg dyspnea score was assessed immediately following the 6-minute walk test. Scores ranged from 0 (for no shortness of breath) to 10 (for greatest shortness of breath ever experienced).
Time Frame: Baseline and Week 12
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | UT-15C (Oral Treprostinil)
Number analyzed (Participants) | 77 | 151
units on a scale
  Borg dyspnea score at Baseline | 3 [2 to 6] | 3 [2 to 4]
  Borg dyspnea score at Week 12 | 3 [2 to 5] | 3 [1 to 5]
  Change in Borg dyspnea score from Baseline to Wk12 | 0 [-1 to 1] | 0 [-1 to 1]
Statistical Analysis 1: Comparison: Placebo vs UT-15C (Oral Treprostinil); Test type: Superiority or Other; p = 0.4887, Wilcoxon rank-sum test; Hodges-Lehmann (H-L) = 0, 95% CI 2-sided [-1 to 0]

8. Secondary Outcome: Dyspnea-Fatigue Index
Description: The dyspnea-fatigue index has three components, each rated on a scale of 0 to 4, for the magnitude of the task that evokes dyspnea or fatigue, the magnitude of the pace (or effort) with which the task is performed and the associated functional impairment in general activities. The ratings for each component were added to form an aggregate score, which could range from 0, for the worst condition, to 12, for the best.
Time Frame: Baseline and Week 12
Population: Two subjects (one in the placebo arm and one in the oral treprostinil arm) from the primary analysis population (n=228) did not have a Baseline dyspnea-fatigue index score and were not included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | UT-15C (Oral Treprostinil)
Number analyzed (Participants) | 76 | 150
units on a scale
  Dyspnea-fatigue index at Baseline | 5.8 (2.4) | 6.2 (2.1)
  Dyspnea-fatigue index at Week 12 | 5.5 (2.9) | 5.9 (2.8)
  Change in dyspnea-fatigue index from BL to Wk 12 | -0.3 (2.5) | -0.3 (2.4)
Statistical Analysis 1: Comparison: Placebo vs UT-15C (Oral Treprostinil); Test type: Superiority or Other; p = 0.6116, Wilcoxon sum-rank test; Hodges-Lehmann (H-L) = 0, 95% CI 2-sided [0 to 1]

9. Secondary Outcome: Symptoms of PAH
Description: Defined symptoms of PAH including fatigue, dyspnea, edema, dizziness, syncope, chest pain, and orthopnea were assessed at Baseline prior to starting study drug and during the Treatment Phase at Week 12. Severity grade values (i.e., 0, 1, 2, or 3 in increasing severity) were assigned for each symptom.
Time Frame: Baseline and Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | UT-15C (Oral Treprostinil)
Number analyzed (Participants) | 77 | 151
units on a scale
  Change in fatigue symptoms | 0.1 (1.0) | 0.0 (1.0)
  Change in dyspnea symptoms | -0.1 (0.9) | -0.2 (0.9)
  Change in edema symptoms | 0.3 (1.0) | 0.2 (1.1)
  Change in dizziness symptoms | 0.0 (1.0) | 0.3 (1.0)
  Change in syncope symptoms | 0.3 (1.0) | 0.3 (0.9)
  Change in chest pain symptoms | 0.1 (0.9) | 0.2 (1.0)
  Change in orthopnea symptoms | 0.2 (0.9) | 0.2 (1.0)

10. Post Hoc Outcome: Six Minute Walk Distance by Baseline WHO Functional Classification III or IV
Description: Exploratory efficacy analyses were to determine the effect of Baseline WHO functional class on treatment effect for change in 6MWD.
  The Hodges-Lehmann median difference between treatment groups was used to estimate the treatment effect on 6MWD from Baseline to Week 12. A rank-based methodology was used instead of parametric-based methodology to avoid statistical bias caused by extreme outliers resulting from the handling of data that are missing due to death or clinical worsening of PAH. It is a more robust estimator than the between-treatment difference in medians.
Time Frame: Baseline and Week 12
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | Placebo | UT-15C (Oral Treprostinil)
Number analyzed (Participants) | 52 | 98
meters
  6MWD at Baseline | 333.5 [269 to 382.5] | 330 [265 to 378]
  6MWD at Week 12 | 316.5 [231.5 to 385] | 354 [265 to 400]
  Change in 6MWD from Baseline to Week 12 | -8.5 [-50.5 to 40] | 20.5 [-20 to 63]
Statistical Analysis 1: Comparison: Placebo vs UT-15C (Oral Treprostinil); Test type: Superiority or Other; p = 0.0326, ANCOVA; Hodges-Lehmann (H-L) = 26, 95% CI 2-sided [1 to 49]

11. Post Hoc Outcome: Six Minute Walk Distance by Baseline WHO Functional Classification: I or II
Description: as for outcome 10
Time Frame: Baseline and Week 12
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | Placebo | UT-15C (Oral Treprostinil)
Number analyzed (Participants) | 25 | 53
meters
  6MWD at Baseline | 370 [297 to 378] | 366 [315 to 390]
  6MWD at Week 12 | 379 [274 to 429] | 391 [348 to 431]
  Change in 6MWD from Baseline to Week 12 | 18 [-30 to 55] | 27 [-5 to 67]
Statistical Analysis 1: Comparison: Placebo vs UT-15C (Oral Treprostinil); Test type: Superiority or Other; p = 0.2275, ANCOVA; Hodges-Lehmann (H-L) = 16.0, 95% CI 2-sided [-15 to 47]

12. Post Hoc Outcome: Six Minute Walk Distance (6MWD) by PAH Etiology: Idiopathic or Heritable PAH
Description: Exploratory efficacy analyses were to determine the effect of PAH etiology (idiopathic/heritable, associated with collagen vascular disease, and other etiologies) on treatment effect for change in 6MWD.
  The Hodges-Lehmann median difference between treatment groups was used to estimate the treatment effect on 6MWD from Baseline to Week 12. A rank-based methodology was used instead of parametric-based methodology to avoid statistical bias caused by extreme outliers resulting from the handling of data that are missing due to death or clinical worsening of PAH. It is a more robust estimator than the between-treatment difference in medians.
Time Frame: Baseline and Week 12
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | Placebo | UT-15C (Oral Treprostinil)
Number analyzed (Participants) | 56 | 114
meters
  6MWD at Baseline | 332.5 [260 to 379] | 346 [281 to 390]
  6MWD at Week 12 | 310.5 [242.5 to 380] | 380 [304 to 420]
  Change in 6MWD from BL to Wk 12 | -7.5 [-50.5 to 42] | 25 [-13 to 67]
Statistical Analysis 1: Comparison: Placebo vs UT-15C (Oral Treprostinil); Test type: Superiority or Other; p = 0.0024, ANCOVA; Hodges-Lehmann (H-L) = 32, 95% CI 2-sided [10 to 55]

13. Post Hoc Outcome: Six Minute Walk Distance (6MWD) for the Entire Study Population
Description: Placebo corrected change in six minute walk distance (6MWD) from Baseline to Week 12, correlates with the historical clinical standard for assessing patient functional status in the treatment of PAH and is considered an objective measure of patient functional status by the American Thoracic Society (ATS). This outcome measure was assessed using data collected from all subjects enrolled in the study, regardless of tablet strength availability at randomization.
  The six minute walk test was to be conducted 3 to 6 house after the previous dose of study drug.
  The Hodges-Lehmann median difference between treatment groups was used to estimate the treatment effect on 6MWD from Baseline to Wk 12. A rank-based methodology was used instead of parametric-based methodology to avoid statistical bias caused by extreme outliers resulting from the handling of data that are missing due to death or clinical worsening of PAH. It is a more robust estimator than the between-treatment difference i
Time Frame: Baseline and Week 12
Population: This analysis was performed using data from all subjects enrolled in the study, regardless of tablet strength availability at randomization.
Measure: Median (Inter-Quartile Range); unit: meters
Groups:
- Placebo: These subjects were randomly allocated to receive placebo twice daily.
- UT-15C (Oral Treprostinil): These subjects were randomly allocated to receive oral treprostinil twice daily.
Arm/Group | Placebo | UT-15C (Oral Treprostinil)
Number analyzed (Participants) | 116 | 233
meters
  6MWD at Baseline | 338.5 [265.5 to 383.5] | 347 [288 to 387]
  6MWD at Week 12 | 329.5 [231.5 to 397.5] | 370 [304 to 420]
  Change in 6MWD from Baseline to Week 12 | 0 [-46 to 40] | 25 [-12 to 63]
Statistical Analysis 1: Comparison: Placebo vs UT-15C (Oral Treprostinil); Test type: Superiority or Other; p = 0.0001, ANCOVA; Hodges-Lehmann (H-L) = 25.5, 95% CI 2-sided [10 to 41]

14. Post Hoc Outcome: Six Minute Walk Distance (6MWD) for the Entire Study Population
Description: Placebo corrected change in six minute walk distance (6MWD) from Baseline to Week 11, a time expected to correlate with trough treprostinil concentration. This outcome measure was assessed using data from all subjects enrolled in the study, regardless of tablet strength availability at the time of randomization.
  The six minute walk test was to be conducted 8 to 13 hours after the previous dose of study drug.
  The Hodges-Lehmann median difference between treatment groups was used to estimate the treatment effect on 6MWD from Baseline to Week 11. A rank-based methodology was used instead of parametric-based methodology to avoid statistical bias caused by extreme outliers resulting from the handling of data that are missing due to death or clinical worsening of PAH. It is a more robust estimator than the between-treatment difference in medians.
Time Frame: Baseline and Week 11
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | Placebo | UT-15C (Oral Treprostinil)
Number analyzed (Participants) | 116 | 233
meters
  6MWD at Baseline | 338.5 [265.5 to 383.5] | 347 [288 to 387]
  6MWD at Week 11 | 326.5 [206 to 398] | 351 [303 to 403]
  Change in 6MWD from Baseline to Week 11 | -2 [-58.5 to 36] | 6 [-18 to 48]
Statistical Analysis 1: Comparison: Placebo vs UT-15C (Oral Treprostinil); Test type: Superiority or Other; p = 0.0025, ANCOVA; Hodges-Lehmann (H-L) = 17, 95% CI 2-sided [3 to 33]

15. Post Hoc Outcome: Six Minute Walk Distance (6MWD) for the Entire Study Population
Description: Placebo corrected change in six minute walk distance (6MWD) from Baseline to Week 8, correlates with the historical clinical standard for assessing patient functional status in the treatment of PAH and is considered an objective measure of patient functional status by the American Thoracic Society (ATS). This outcome measure was assessed using data from all subjects enrolled in the study, regardless of tablet strength availability at randomization.
  The six minute walk test was to be conducted 3 to 6 house after the previous dose of study drug.
  The Hodges-Lehmann median difference between treatment groups was used to estimate the treatment effect on 6MWD from Baseline to Week 8. A rank-based methodology was used instead of parametric-based methodology to avoid statistical bias caused by extreme outliers resulting from the handling of data that are missing due to death or clinical worsening of PAH. It is a more robust estimator than the between-treatment difference in medians.
Time Frame: Baseline and Week 8
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | Placebo | UT-15C (Oral Treprostinil)
Number analyzed (Participants) | 116 | 233
meters
  6MWD at Baseline | 338.5 [265.5 to 383.5] | 347 [288 to 387]
  6MWD at Week 8 | 339.5 [227 to 392] | 360 [300 to 411]
  Change in 6MWD from Baseline to Week 8 | 1.0 [-38.5 to 34.5] | 17.0 [-13 to 54]
Statistical Analysis 1: Comparison: Placebo vs UT-15C (Oral Treprostinil); Test type: Superiority or Other; p = 0.0008, ANCOVA; Hodges-Lehmann (H-L) = 20, 95% CI 2-sided [7 to 34]

16. Post Hoc Outcome: Six Minute Walk Distance (6MWD) for the Entire Study Population
Description: Placebo corrected change in six minute walk distance (6MWD) from Baseline to Week 4, correlates with the historical clinical standard for assessing patient functional status in the treatment of PAH and is considered an objective measure of patient functional status by the American Thoracic Society (ATS). This outcome measure was assessed using data from all subjects enrolled in the study, regardless of tablet strength availability at randomization.
  The six minute walk test was to be conducted 3 to 6 house after the previous dose of study drug.
  The Hodges-Lehmann median difference between treatment groups was used to estimate the treatment effect on 6MWD from Baseline to Week 4. A rank-based methodology was used instead of parametric-based methodology to avoid statistical bias caused by extreme outliers resulting from the handling of data that are missing due to death or clinical worsening of PAH. It is a more robust estimator than the between-treatment difference in medians.
Time Frame: Baseline and Week 4
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | Placebo | UT-15C (Oral Treprostinil)
Number analyzed (Participants) | 116 | 233
meters
  6MWD at Baseline | 338.5 [265.5 to 383.5] | 347 [288 to 387]
  6MWD at Week 4 | 339.5 [251 to 387] | 358 [288 to 403.2]
  Change in 6MWD from Baseline to Week 4 | -4 [-31.5 to 20] | 7 [-13 to 42]
Statistical Analysis 1: Comparison: Placebo vs UT-15C (Oral Treprostinil); Test type: Superiority or Other; p = 0.0025, ANCOVA; Hodges-Lehmann (H-L) = 14, 95% CI 2-sided [3.9 to 25]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded throughout the 12 week study which was conducted between October 2006 and April 2011.
Description: Adverse events are reported for the modified intention to treat (mITT) group, which includes subjects with access to 0.25 mg tablets at randomization (n=228).
Arm/Group | Placebo | UT-15C (Oral Treprostinil)
All-Cause Mortality (participants affected / at risk) | 6/77 | 9/151
Serious Adverse Events (participants affected / at risk) | 15/77 | 27/151
Other Adverse Events (participants affected / at risk) | 68/77 | 138/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=77) | UT-15C (Oral Treprostinil) (N=151)
right ventricular failure (Cardiac disorders) | 3 (3) | 10 (12)
pulmonary hypertension (Cardiac disorders) | 4 (4) | 3 (3)
death (General disorders) | 2 (2) | 2 (2)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
anterograde amnesia (Nervous system disorders) | 0 (0) | 1 (1)
cardiac failure (Cardiac disorders) | 0 (0) | 1 (2)
cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
circulatory collapse (Cardiac disorders) | 1 (1) | 0 (0)
collagen-vascular disease (Vascular disorders) | 1 (1) | 0 (0)
cor pulmonale acute (Cardiac disorders) | 0 (0) | 1 (1)
diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
diarrhea infectious (Gastrointestinal disorders) | 1 (1) | 0 (0)
paroxysmal noturnal dypsnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 0 (0) | 1 (1)
lower respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
palpitations (Cardiac disorders) | 1 (1) | 0 (0)
presyncope (General disorders) | 0 (0) | 1 (1)
pulmonary edema (Cardiac disorders) | 0 (0) | 1 (1)
acute renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
septic shock (Infections and infestations) | 0 (0) | 1 (1)
skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
sudden death (General disorders) | 0 (0) | 1 (1)
syncope (General disorders) | 0 (0) | 1 (1)
systemic lupus erythematosus (Immune system disorders) | 0 (0) | 1 (1)
urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
sudden cardiac death (Cardiac disorders) | 0 (0) | 1 (1)
renal impairment (Renal and urinary disorders) | 0 (0) | 1 (2)
respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=77) | UT-15C (Oral Treprostinil) (N=151)
headache (Nervous system disorders) | 15 (17) | 95 (131)
diarrhea (Gastrointestinal disorders) | 12 (12) | 46 (54)
nausea (Gastrointestinal disorders) | 14 (14) | 45 (50)
vomiting (Gastrointestinal disorders) | 12 (12) | 26 (31)
flushing (Vascular disorders) | 5 (5) | 23 (25)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6) | 21 (25)
pain in jaw (Musculoskeletal and connective tissue disorders) | 3 (3) | 17 (18)
fatigue (General disorders) | 6 (6) | 14 (15)
abdominal pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 13 (13)
peripheral edema (Vascular disorders) | 5 (5) | 13 (15)
hypokalemia (Endocrine disorders) | 2 (3) | 13 (16)
decreased appetite (General disorders) | 4 (4) | 12 (12)
insomnia (Nervous system disorders) | 2 (2) | 11 (12)
right ventricular failure (Cardiac disorders) | 3 (3) | 10 (12)
nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 9 (12)
abdominal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 9 (9)
upper abdominal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 8 (12)
back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 7 (8)
arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 7 (7)
gastritis (Gastrointestinal disorders) | 1 (1) | 7 (7)
pain (General disorders) | 0 (0) | 7 (7)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 7 (7)
asthenia (General disorders) | 4 (4) | 6 (9)
muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (8)
pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
oropharyngeal pain (General disorders) | 4 (4) | 1 (1)
dizziness (General disorders) | 11 (11) | 17 (19)
pyrexia (Infections and infestations) | 8 (8) | 7 (7)
upper respiratory tract infection (Infections and infestations) | 5 (5) | 8 (8)
cough (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 14 (15)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the results of this trial must be consistent with the United Therapeutics publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.